CLINICAL TRIAL: NCT03813056
Title: A Phase II, Interventional, Double-blind, Single-center Study of the Effects of Ripasudil on Cornea Clearing After Descemet Membrane Endothelial Keratoplasty in Subjects With Fuchs' Endothelial Corneal Dystrophy
Brief Title: Ripasudil for Enhanced Corneal Clearing Following Descemet Membrane Endothelial Keratoplasty in Fuchs' Dystrophy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michael D. Straiko, MD (Other)
Collaborators: Lions VisionGift Research (Other); Eye Bank Association of America (Other)
Responsible Party: Sponsor-Investigator, Michael D. Straiko, MD, Associate Director of Corneal Services, Devers Eye Institute, Legacy Health System
Organization: Legacy Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDMEK-01
Record Dates: First submitted 2019-01-19; First posted 2019-01-23 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Fuchs Endothelial Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy | interventions — K-115; Ophthalmic Solutions; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glanatec (Experimental): Glanatec eye drops will be administered 6x per day for 2-4 weeks
  Interventions: Drug: Glanatec; Procedure: Descemet Membrane Endothelial Keratoplasty
- Placebo Control (Placebo Comparator): Optive artificial tears will be administered 6x per day for 2-4 weeks
  Interventions: Drug: Optive, Ophthalmic Solution; Procedure: Descemet Membrane Endothelial Keratoplasty

INTERVENTIONS:
Drug: Glanatec — Rho kinase Inhibitor
  Other Names: Ripasudil
  Arms: Glanatec
Drug: Optive, Ophthalmic Solution — artificial tears (placebo)
  Other Names: Optive, artificial tears
  Arms: Placebo Control
Procedure: Descemet Membrane Endothelial Keratoplasty — Partial thickness corneal transplant that replaces only the diseased corneal endothelium and descemet membrane of the recipient.
  Other Names: DMEK

SUMMARY:
Recently, published literature has reported that performing a descemetorhexis in combination with topical Rho kinase (ROCK) inhibitor therapy was successful in clearing edematous corneas in patients with Fuchs Endothelial Corneal Dystrophy.

Ripasudil hydrochloride hydrate( Glanatec ophthalmic solution 0.4%), a potent ROCK inhibitor, has been approved in Japan since 2014 for ocular use in the treatment of glaucoma. Ripasudil acts as an IOP-lowering drug by affecting aqueous outflow through the trabecular meshwork and Schlemm's canal.

The goal of this study is to test the potential benefits of Ripasudil therapy administered after Descemet Membrane Endothelial Keratoplasty (DMEK) surgery. We believe that performing a standard DMEK surgery in combination with Ripasudil treatment in patients with Fuchs Endothelial Corneal Dystrophy could accelerate endothelial cell healing and clear edematous corneas faster, with less post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed clinically with Fuchs endothelial corneal dystrophy by the study investigator.
* Phakic or pseudophakic with posterior capsule supported, suture-fixated, or sulcus-supported posterior chamber intraocular lens.
* Fuchs dystrophy grades 2-5 on the Krachmer grading scale.
* Presence of central guttae and/or stromal edema being the primary cause of decreased vision.
* The peripheral cornea to the central 6mm is devoid of guttata changes.
* Best corrected visual acuity in the study eye is 20/40 or worse with glare testing at study enrollment.

Exclusion Criteria:

* Uncontrolled glaucoma (IOP >25 mmHg).
* Presence of secondary corneal pathology such as infective or autoimmune keratitis.
* Advanced corneal stromal edema with bullae on slit-lamp biomicroscopy.
* History of herpes simplex virus or cytomegalovirus keratitis.
* Prior penetrating keratoplasty.
* Aphakic in study eye.
* Allergy to any component of the Ripasudil hydrochloride hydrate 0.4% that will be used in the course of the study.
* Tubes or trabeculectomy from prior glaucoma surgery.

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Time to corneal clearance | 6 months
  Slit lamp examinations and corneal OCT measurements will be taken in a longitudinal fashion to compare corneal clearance and stabilization.

SECONDARY OUTCOMES:
Best corrected visual acuity | 6 months
  Longitudinal best corrected visual acuity tests will be performed to compare the time course of best vision attained and reported in Snellen units.
Endothelial cell density | 6 months
  Specular imaging will be conducted at 3 and 6 month postoperative to compare endothelial cells loss.
Post surgery complications | 6 months
  Number of graft detachments requiring a re-bubble procedure and number of graft failures will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Straiko, M.D., Principal Investigator — Devers Eye Institute
Locations (1):
- Devers Eye Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No